CLINICAL TRIAL: NCT00843089
Title: Secondary Prevention After Coronary Bypass Surgery: A Pilot Study
Brief Title: Secondary Prevention After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Kramer, MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Kramer, MD, CTS SURGEON, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11562
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; CABG
MeSH Terms: conditions — Coronary Artery Disease | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard care
- 2 (Experimental): Educational session with pharmacist, nutritionist, and cardiac rehabilitation nurse
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Educational session with pharmacist, nutritionist, and cardiac rehabilitation nurse
  Arms: 2

SUMMARY:
Despite immediate symptomatic success after coronary bypass surgery in patients with coronary artery disease, this effect is not sustained over time since risk factors for coronary artery disease are still in place. The role of secondary prevention becomes increasingly important as it can potentially decrease or eliminate the need for another intervention in these high risk subjects. This project seeks to evaluate the effect of emphasizing secondary prevention measures in this patient population during hospital admission and through six months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 who will undergo a CABG procedure and who have given written informed consent

Exclusion Criteria:

* Subjects under the age of 18 or who are unable to give consent on their own behald

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
compliance with medications and lifestyle changes | Month 1, 3, 6 and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kramer, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States